CLINICAL TRIAL: NCT06222593
Title: A Phase I/II Study to Evaluate the Safety and Efficacy of Bicalutamide in Combination with Sunitinib in Patients with Receptor Tyrosine Kinase Inhibitor Resistant Renal Cell Carcinoma
Brief Title: Study to Evaluate the Safety and Efficacy of Bicalutamide in Combination with Sunitinib in Patients with TKIs-resistant RCC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Roberto Pili, Chief, Division of Hematology/Oncology, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006224
Record Dates: First submitted 2022-11-11; First posted 2024-01-24 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-09

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — bicalutamide; Sunitinib

STUDY DESIGN:
Intervention Model Description: Longitudinal
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bicalutamide in combination with Sunitinib (Experimental): Bicalutamide 50mg once a day (QD) in combination with sunitinib 37.5mg, 25mg or 50mg QD (2 weeks ON, 1 week OFF). Four or more 21 day-long cycles.
  Interventions: Drug: Bicalutamide in combination with Sunitinib

INTERVENTIONS:
Drug: Bicalutamide in combination with Sunitinib — Antineoplastics, Antiandrogen; CYP3A4 Inhibitor
  Other Names: (RS)-N-[4-cyano-3-(trifluoromethyl)phenyl]-3-[(4-fluorophenyl sulfonyl]-2-hydroxy-2-methylpropanamide; UNII: A0Z3NAU9DP; CASODEX

SUMMARY:
This is a Phase I/II open-label, efficacy and safety study of bicalutamide in combination with sunitinib in patients with advanced renal cell carcinoma (RCC) who have been treated with a receptor tyrosine kinase inhibitor (RTKI) and experienced disease progression.

DETAILED DESCRIPTION:
This is a Phase I/II open-label, efficacy and safety study of bicalutamide in combination with sunitinib in patients with advanced renal cell carcinoma (RCC) who have been treated with a receptor tyrosine kinase inhibitor (RTKI) and experienced disease progression. After entering the study, patients will have sunitinib dosed at the 2 weeks ON and one week OFF scheduled. Dose and schedule modification of sunitinib will be allowed at the discretion of the treating physician. Bicalutamide will be administrated orally at 50 mg daily. This clinical study will utilize the Simon's optimal two stage design. Investigators will enroll 9 patients in the first stage. If no response is seen, then the trial is terminated for futility. Otherwise, accrual continues to a total of 16 patients. If at most 2 patients respond among the 16 patients, this therapy would warrant further investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial.
2. Be greater than or equal to 18 years of age on day of signing informed consent.
3. Have measurable disease based on RECIST 1.1
4. Have a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
5. Demonstrate adequate organ function
6. Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication.
7. Subjects of childbearing potential should be willing to use 2 methods of contraception for the course of the study through 120 days after the last dose of study medication
8. Male subjects without a previous vasectomy should agree to use an adequate method of contraception (i.e. abstinence, condom with spermicidal foam/gel/film/cream) starting with the first dose of study therapy through 120 days after the last dose of study therapy.
9. Subjects have archival tumor tissue available or are willing to undergo a baseline biopsy prior to treatment.
10. Subjects must have a life expectancy of at least 6 months.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has active Bacillus tuberculosis (TB)
4. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
5. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
6. Has an active infection requiring systemic therapy.
7. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
8. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
9. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
10. Has a known history of Human Immunodeficiency Virus (HIV)
11. Has known active Hepatitis B or Hepatitis C
12. Has received a live vaccine within 30 days of planned start of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
To assess safety and tolerability of bicalutamide in combination with sunitinib in patients with RTKIs-resistant renal cell carcinoma. | 3 years
  Investigators will report the number of participants with treatment-related adverse events as assessed by CTCAE v4.0.
To assess efficacy of bicalutamide in combination with sunitinib in patients with RTKIs-resistant renal cell carcinoma. | 3 years
  Investigators will also report the number of patients who achieve either partial or complete response by RECIST criteria on tumor imaging.

OTHER OUTCOMES:
To characterize androgen receptor (AR) expression in tumor samples immunohistochemistry (IHC) | 3 years
  The outcome measure is IHC score (scale goes from 0-3, 0 being better outcome and 3 being the worst outcome) (0): negative staining
  1. : weak staining
  2. : moderate staining
  3. : strong staining
To characterize expression of AR-related micro-RNA (miR) in tumor and/or blood by polymerase chain reaction (PCR) | 3 years
  Outcome measure: ratio of miR expression with respect to the gene of reference
To characterize Kallikrein-2 (KLK2) expression in blood by ELISA | 3 years
  ELISA test calculates the concentration of protein as ng per ml of serum/blood.
To characterize KLK2 expression in tumor samples immunohistochemistry (IHC) | 3 years
  The outcome measure is IHC score (scale goes from 0-3, 0 being better outcome and 3 being the worst outcome) (0): negative staining
  1. : weak staining
  2. : moderate staining
  3. : strong staining

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Pili, MD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- UB/ Great Lakes Cancer Care, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No